CLINICAL TRIAL: NCT06588270
Title: Effect of Virtual Reality-based Therapy on Negative Symptoms in People with Schizophrenia: Study Protocol for a Randomized Controlled Trial
Brief Title: Effect of Virtual Reality-based Therapy on Negative Symptoms in People with Schizophrenia
Acronym: VR-SCHIZO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de la Florida Dra. Eloiza Diaz (Other)
Responsible Party: Principal Investigator, Javiera Libuy Mena, Director, Hospital de la Florida Dra. Eloiza Diaz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA20I0002; SA20I0002 (Other Grant/Funding Number: Agencia Nacional de Investigación y Desarrollo, Chile)
Record Dates: First submitted 2022-11-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Virtual reality; Negative symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: The study will be a double-blind, randomized controlled trial (RCT). Patients will be divided into two groups. The intervention group will receive a VR experience with a treatment software, while the control group will receive a VR experience without the software. All patients will continue on their current medications
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of allocation will be maintained for the research workers until all outcome measures for all participants have been collected. Blindness will be maintained using a range of measures (e.g. separate offices for therapist and researchers, protocols for answering phones and emails and security for electronic randomization information). The trial statistician will be also blind to the randomization outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality-based therapy (Experimental): The intervention group will receive a VR experience with a treatment software. The aim is to immerse the patient in an interactive environment that invites him/her to explore and complete goal-directed activities with sensory, visual and/or auditory rewards.
  The therapy will be delivered with the support of a therapist once per week for 12 consecutive weeks. Each therapy session will last approximately 20 minutes.
  Interventions: Behavioral: Virtual Reality Therapy for the Negative Symptoms of Schizophrenia
- Sham -VR (Sham Comparator): Control group's patients will continue pharmacological and non pharmacological usual treatment. Additionally, these patients will attend to VR sessions without the software created activities for treatment (sham-VR). Sessions will be the same length and quantity as the intervention group's sessions.
  Interventions: Behavioral: Sham- VR

INTERVENTIONS:
Behavioral: Virtual Reality Therapy for the Negative Symptoms of Schizophrenia — VRTNSS is a 12-session therapy using psychological intervention principles. Each therapy session will involve engaging with different VR based tasks where participants can experience different activities.
  Arms: Virtual reality-based therapy
Behavioral: Sham- VR — Patients will attend to VR sessions without the software created activities for treatment (sham-VR).
  Arms: Sham -VR

SUMMARY:
A randomised, controlled, double-blind clinical trial will be carried out to evaluate the effectiveness of a VR assisted treatment for negative symptoms in people with schizophrenia. Patients with a standardised diagnosis of schizophrenia meeting the inclusion criteria will receive 12 weekly sessions of VR assisted therapy plus treatment as usual (TAU). A control group will be exposed to a neutral VR environment plus TAU. The hypothesis is that patients who are treated with active VR assisted therapy will have less negative symptoms as rated by the PANSS-N scale, compared to the control group.

The protocol was approved by the hospital ethics committee of the Servicio de Salud Metropolitano Suroriente. Patients sign an informed consent form, from which they may withdraw at any point during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia made by the treating psychiatrist and corroborated by a team's psychiatrist under CIE-10 criteria.
* Age between 18 to 65 years-old.
* Outpatient setting,
* Clinical stability defined as no psychiatric hospitalizations in the last 6 months and not currently on queue for psychiatric hospitalization.
* No concomitant active substance abuse disorder, excluding nicotine.
* Subjects are capable of providing informed consent.

Exclusion Criteria:

* Previous diagnosis of learning disability according either to ICD- 10 or clinical history
* Verbal expression difficulties, determined by language or medical causes.
* Deafness and/or blindness.
* Other physical handicaps to use VR devices.
* Predominant positive symptoms, defined as PANNS-C > 0.
* Catatonic symptoms.
* Previous epilepsy diagnosis.
* Neurodegenerative disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Negative symptoms | 12 weeks
  The primary outcome will be the difference in the rate of change in negative symptoms at 3 months of follow-up. Negative symptoms are measured with the Positive and negative syndrome scale (PANSS) negative subscale. Scale's scoring system ranges from 7 to 49 points.
  A 25% reduction from the baseline score on the PANSS-N will be considered a significant decrease.

SECONDARY OUTCOMES:
Positive symptoms | 12 weeks
  Positive symptoms are measured with the Positive and negative syndrome scale (PANSS) positive subscale. It consists of seven items: delusions, conceptual disorganization, hallucinations, excitement, grandiosity, suspiciousness/persecution and hostility. Scale's scoring system ranges from 7 to 49 points. No changes from the baseline PANSS-P score are expected.
Mood symptoms | 12 weeks
  Mood symptoms are assessed with the Calgary depression scale for schizophrenia. Scale's scoring system ranges from 0 to 27 points.
Quality of life: Short Form (36) Health Survey | 12 weeks
  The Short Form (36) Health Survey is a self-applied questionnaire that addresses eight life dimensions: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. It will be used to assess quality of life. As it is a dimensional scale, it does not have a cutoff score.
Global functioning | 12 weeks
  Global assessment of functioning (GAF) is a numeric scale of social, occupational and psychological functioning. Scale's scoring system ranges from 10 to 100 points.
Social anxiety | 12 weeks
  Social anxiety symptoms are measured with Social Interaction Anxiety Scale (SIAS). This is a self applied, twenty items instrument. Scale's scoring system ranges from 0 to 80 points.
Adverse effects | 12 weeks
  Adverse effects are measured with the Simulator Sickness Questionnaire (SSQ). This instrument assesses 16 subjective items and was developed to accommodate symptoms specific to simulator technology. It can be self applied or clinician rated. Participants are asked to assign a score from 0-3 for each of the sixteen items on the SSQ. Total scores can be associated with negligible (< 5), minimal (5 - 10), significant (10 - 15), concerning (15 - 20) and bad (>20) symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico La Florida, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Saha S, Chant D, Welham J, McGrath J. A systematic review of the prevalence of schizophrenia. PLoS Med. 2005 May;2(5):e141. doi: 10.1371/journal.pmed.0020141. Epub 2005 May 31. PMID 15916472
- [Background] McGrath J, Saha S, Chant D, Welham J. Schizophrenia: a concise overview of incidence, prevalence, and mortality. Epidemiol Rev. 2008;30:67-76. doi: 10.1093/epirev/mxn001. Epub 2008 May 14. PMID 18480098
- [Background] Vicente B, Rioseco P, Saldivia S, Kohn R, Torres S. [Chilean study on the prevalence of psychiatric disorders (DSM-III-R/CIDI) (ECPP)]. Rev Med Chil. 2002 May;130(5):527-36. Spanish. PMID 12143273
- [Background] Gonzalez-Valderrama A, Jongsma HE, Mena C, Castaneda CP, Nachar R, Undurraga J, Crossley N, Aceituno D, Iruretagoyena B, Gallardo C, Mondaca P, Monje M, Irarrazaval M, Zavala C, Valmaggia L, Kirkbride JB. The incidence of non-affective psychotic disorders in Chile between 2005 and 2018: results from a national register of over 30 000 cases. Psychol Med. 2022 Apr;52(5):914-923. doi: 10.1017/S0033291720002664. Epub 2020 Aug 6. PMID 32758314
- [Background] GBD 2019 Mental Disorders Collaborators. Global, regional, and national burden of 12 mental disorders in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Psychiatry. 2022 Feb;9(2):137-150. doi: 10.1016/S2215-0366(21)00395-3. Epub 2022 Jan 10. PMID 35026139
- [Background] Cloutier M, Aigbogun MS, Guerin A, Nitulescu R, Ramanakumar AV, Kamat SA, DeLucia M, Duffy R, Legacy SN, Henderson C, Francois C, Wu E. The Economic Burden of Schizophrenia in the United States in 2013. J Clin Psychiatry. 2016 Jun;77(6):764-71. doi: 10.4088/JCP.15m10278. PMID 27135986
- [Background] Hjorthoj C, Sturup AE, McGrath JJ, Nordentoft M. Years of potential life lost and life expectancy in schizophrenia: a systematic review and meta-analysis. Lancet Psychiatry. 2017 Apr;4(4):295-301. doi: 10.1016/S2215-0366(17)30078-0. Epub 2017 Feb 22. PMID 28237639
- [Background] Saha S, Chant D, McGrath J. A systematic review of mortality in schizophrenia: is the differential mortality gap worsening over time? Arch Gen Psychiatry. 2007 Oct;64(10):1123-31. doi: 10.1001/archpsyc.64.10.1123. PMID 17909124
- [Background] Avila C, Holloway AC, Hahn MK, Morrison KM, Restivo M, Anglin R, Taylor VH. An Overview of Links Between Obesity and Mental Health. Curr Obes Rep. 2015 Sep;4(3):303-10. doi: 10.1007/s13679-015-0164-9. PMID 26627487
- [Background] Harvey PD, Strassnig M. Predicting the severity of everyday functional disability in people with schizophrenia: cognitive deficits, functional capacity, symptoms, and health status. World Psychiatry. 2012 Jun;11(2):73-9. doi: 10.1016/j.wpsyc.2012.05.004. PMID 22654932
- [Background] Galderisi S, Rossi A, Rocca P, Bertolino A, Mucci A, Bucci P, Rucci P, Gibertoni D, Aguglia E, Amore M, Bellomo A, Biondi M, Brugnoli R, Dell'Osso L, De Ronchi D, Di Emidio G, Di Giannantonio M, Fagiolini A, Marchesi C, Monteleone P, Oldani L, Pinna F, Roncone R, Sacchetti E, Santonastaso P, Siracusano A, Vita A, Zeppegno P, Maj M; Italian Network For Research on Psychoses. The influence of illness-related variables, personal resources and context-related factors on real-life functioning of people with schizophrenia. World Psychiatry. 2014 Oct;13(3):275-87. doi: 10.1002/wps.20167. PMID 25273301
- [Background] Rabinowitz J, Levine SZ, Garibaldi G, Bugarski-Kirola D, Berardo CG, Kapur S. Negative symptoms have greater impact on functioning than positive symptoms in schizophrenia: analysis of CATIE data. Schizophr Res. 2012 May;137(1-3):147-50. doi: 10.1016/j.schres.2012.01.015. Epub 2012 Feb 6. PMID 22316568
- [Background] Jauhar S, McKenna PJ, Radua J, Fung E, Salvador R, Laws KR. Cognitive-behavioural therapy for the symptoms of schizophrenia: systematic review and meta-analysis with examination of potential bias. Br J Psychiatry. 2014 Jan;204(1):20-9. doi: 10.1192/bjp.bp.112.116285. PMID 24385461
- [Background] McCutcheon RA, Pillinger T, Mizuno Y, Montgomery A, Pandian H, Vano L, Marques TR, Howes OD. The efficacy and heterogeneity of antipsychotic response in schizophrenia: A meta-analysis. Mol Psychiatry. 2021 Apr;26(4):1310-1320. doi: 10.1038/s41380-019-0502-5. Epub 2019 Aug 30. PMID 31471576
- [Background] Galderisi S, Mucci A, Buchanan RW, Arango C. Negative symptoms of schizophrenia: new developments and unanswered research questions. Lancet Psychiatry. 2018 Aug;5(8):664-677. doi: 10.1016/S2215-0366(18)30050-6. Epub 2018 Mar 27. PMID 29602739
- [Background] Fusar-Poli P, Papanastasiou E, Stahl D, Rocchetti M, Carpenter W, Shergill S, McGuire P. Treatments of Negative Symptoms in Schizophrenia: Meta-Analysis of 168 Randomized Placebo-Controlled Trials. Schizophr Bull. 2015 Jul;41(4):892-9. doi: 10.1093/schbul/sbu170. Epub 2014 Dec 20. PMID 25528757
- [Background] Kahn RS, Sommer IE, Murray RM, Meyer-Lindenberg A, Weinberger DR, Cannon TD, O'Donovan M, Correll CU, Kane JM, van Os J, Insel TR. Schizophrenia. Nat Rev Dis Primers. 2015 Nov 12;1:15067. doi: 10.1038/nrdp.2015.67. PMID 27189524
- [Background] Jaaskelainen E, Juola P, Hirvonen N, McGrath JJ, Saha S, Isohanni M, Veijola J, Miettunen J. A systematic review and meta-analysis of recovery in schizophrenia. Schizophr Bull. 2013 Nov;39(6):1296-306. doi: 10.1093/schbul/sbs130. Epub 2012 Nov 20. PMID 23172003
- [Background] Rus-Calafell M, Garety P, Sason E, Craig TJK, Valmaggia LR. Virtual reality in the assessment and treatment of psychosis: a systematic review of its utility, acceptability and effectiveness. Psychol Med. 2018 Feb;48(3):362-391. doi: 10.1017/S0033291717001945. Epub 2017 Jul 24. PMID 28735593
- [Background] Strickland D. Virtual reality for the treatment of autism. Stud Health Technol Inform. 1997;44:81-6. PMID 10184809
- [Background] Valmaggia LR, Freeman D, Green C, Garety P, Swapp D, Antley A, Prescott C, Fowler D, Kuipers E, Bebbington P, Slater M, Broome M, McGuire PK. Virtual reality and paranoid ideations in people with an 'at-risk mental state' for psychosis. Br J Psychiatry Suppl. 2007 Dec;51:s63-8. doi: 10.1192/bjp.191.51.s63. PMID 18055940
- [Background] da Costa RM, de Carvalho LA. The acceptance of virtual reality devices for cognitive rehabilitation: a report of positive results with schizophrenia. Comput Methods Programs Biomed. 2004 Mar;73(3):173-82. doi: 10.1016/S0169-2607(03)00066-X. PMID 14980398
- [Background] Fornells-Ambrojo M, Barker C, Swapp D, Slater M, Antley A, Freeman D. Virtual reality and persecutory delusions: safety and feasibility. Schizophr Res. 2008 Sep;104(1-3):228-36. doi: 10.1016/j.schres.2008.05.013. Epub 2008 Jun 24. PMID 18571899
- [Background] Ku J, Jang HJ, Kim KU, Park SH, Kim JJ, Kim CH, Nam SW, Kim IY, Kim SI. Pilot study for assessing the behaviors of patients with schizophrenia towards a virtual avatar. Cyberpsychol Behav. 2006 Oct;9(5):531-9. doi: 10.1089/cpb.2006.9.531. PMID 17034319
- [Background] Wilkins LK, Girard TA, King J, King MJ, Herdman KA, Christensen BK, King J. Spatial-memory deficit in schizophrenia spectrum disorders under viewpoint-independent demands in the virtual courtyard task. J Clin Exp Neuropsychol. 2013;35(10):1082-93. doi: 10.1080/13803395.2013.857389. Epub 2013 Nov 13. PMID 24219234
- [Background] Wilkins LK, Girard TA, Konishi K, King M, Herdman KA, King J, Christensen B, Bohbot VD. Selective deficit in spatial memory strategies contrast to intact response strategies in patients with schizophrenia spectrum disorders tested in a virtual navigation task. Hippocampus. 2013 Nov;23(11):1015-24. doi: 10.1002/hipo.22189. PMID 23939937
- [Background] Sorkin A, Weinshall D, Modai I, Peled A. Improving the accuracy of the diagnosis of schizophrenia by means of virtual reality. Am J Psychiatry. 2006 Mar;163(3):512-20. doi: 10.1176/appi.ajp.163.3.512. PMID 16513875
- [Background] Sorkin A, Weinshall D, Peled A. The distortion of reality perception in schizophrenia patients, as measured in Virtual Reality. Stud Health Technol Inform. 2008;132:475-80. PMID 18391348
- [Background] Weniger G, Irle E. Allocentric memory impaired and egocentric memory intact as assessed by virtual reality in recent-onset schizophrenia. Schizophr Res. 2008 Apr;101(1-3):201-9. doi: 10.1016/j.schres.2008.01.011. Epub 2008 Feb 13. PMID 18276116
- [Background] Fajnerova I, Rodriguez M, Levcik D, Konradova L, Mikolas P, Brom C, Stuchlik A, Vlcek K, Horacek J. A virtual reality task based on animal research - spatial learning and memory in patients after the first episode of schizophrenia. Front Behav Neurosci. 2014 May 27;8:157. doi: 10.3389/fnbeh.2014.00157. eCollection 2014. PMID 24904329
- [Background] Josman N, Schenirderman AE, Klinger E, Shevil E. Using virtual reality to evaluate executive functioning among persons with schizophrenia: a validity study. Schizophr Res. 2009 Dec;115(2-3):270-7. doi: 10.1016/j.schres.2009.09.015. Epub 2009 Oct 22. PMID 19850451
- [Background] Synofzik M, Thier P, Leube DT, Schlotterbeck P, Lindner A. Misattributions of agency in schizophrenia are based on imprecise predictions about the sensory consequences of one's actions. Brain. 2010 Jan;133(Pt 1):262-71. doi: 10.1093/brain/awp291. Epub 2009 Dec 7. PMID 19995870
- [Background] Landgraf S, Krebs MO, Olie JP, Committeri G, van der Meer E, Berthoz A, Amado I. Real world referencing and schizophrenia: are we experiencing the same reality? Neuropsychologia. 2010 Aug;48(10):2922-30. doi: 10.1016/j.neuropsychologia.2010.05.034. Epub 2010 Jun 9. PMID 20540956
- [Background] Kurtz MM, Baker E, Pearlson GD, Astur RS. A virtual reality apartment as a measure of medication management skills in patients with schizophrenia: a pilot study. Schizophr Bull. 2007 Sep;33(5):1162-70. doi: 10.1093/schbul/sbl039. Epub 2006 Sep 6. PMID 16956984
- [Background] Craig TK, Rus-Calafell M, Ward T, Leff JP, Huckvale M, Howarth E, Emsley R, Garety PA. AVATAR therapy for auditory verbal hallucinations in people with psychosis: a single-blind, randomised controlled trial. Lancet Psychiatry. 2018 Jan;5(1):31-40. doi: 10.1016/S2215-0366(17)30427-3. Epub 2017 Nov 23. PMID 29175276
- [Background] Percie du Sert O, Potvin S, Lipp O, Dellazizzo L, Laurelli M, Breton R, Lalonde P, Phraxayavong K, O'Connor K, Pelletier JF, Boukhalfi T, Renaud P, Dumais A. Virtual reality therapy for refractory auditory verbal hallucinations in schizophrenia: A pilot clinical trial. Schizophr Res. 2018 Jul;197:176-181. doi: 10.1016/j.schres.2018.02.031. Epub 2018 Feb 24. PMID 29486956
- [Background] Leff J, Williams G, Huckvale MA, Arbuthnot M, Leff AP. Computer-assisted therapy for medication-resistant auditory hallucinations: proof-of-concept study. Br J Psychiatry. 2013 Jun;202:428-33. doi: 10.1192/bjp.bp.112.124883. Epub 2013 Feb 21. PMID 23429202
- [Background] Freeman D, Bradley J, Antley A, Bourke E, DeWeever N, Evans N, Cernis E, Sheaves B, Waite F, Dunn G, Slater M, Clark DM. Virtual reality in the treatment of persecutory delusions: randomised controlled experimental study testing how to reduce delusional conviction. Br J Psychiatry. 2016 Jul;209(1):62-7. doi: 10.1192/bjp.bp.115.176438. Epub 2016 May 5. PMID 27151071
- [Background] Gega L, White R, Clarke T, Turner R, Fowler D. Virtual environments using video capture for social phobia with psychosis. Cyberpsychol Behav Soc Netw. 2013 Jun;16(6):473-9. doi: 10.1089/cyber.2013.1510. Epub 2013 May 9. PMID 23659722
- [Background] Rus-Calafell M, Gutierrez-Maldonado J, Ribas-Sabate J. A virtual reality-integrated program for improving social skills in patients with schizophrenia: a pilot study. J Behav Ther Exp Psychiatry. 2014 Mar;45(1):81-9. doi: 10.1016/j.jbtep.2013.09.002. Epub 2013 Sep 11. PMID 24063993
- [Background] Park KM, Ku J, Choi SH, Jang HJ, Park JY, Kim SI, Kim JJ. A virtual reality application in role-plays of social skills training for schizophrenia: a randomized, controlled trial. Psychiatry Res. 2011 Sep 30;189(2):166-72. doi: 10.1016/j.psychres.2011.04.003. Epub 2011 Apr 29. PMID 21529970
- [Background] Tsang MM, Man DW. A virtual reality-based vocational training system (VRVTS) for people with schizophrenia in vocational rehabilitation. Schizophr Res. 2013 Mar;144(1-3):51-62. doi: 10.1016/j.schres.2012.12.024. Epub 2013 Jan 26. PMID 23356951
- [Background] Rebenitsch L, Owen C. Review on cybersickness in applications and visual displays. Virtual Reality. 2016. 20:101-12.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Peralta Martin V, Cuesta Zorita MJ. [Validation of positive and negative symptom scale (PANSS) in a sample of Spanish schizophrenic patients]. Actas Luso Esp Neurol Psiquiatr Cienc Afines. 1994 Jul-Aug;22(4):171-7. Spanish. PMID 7810373
- [Background] Addington D, Addington J, Schissel B. A depression rating scale for schizophrenics. Schizophr Res. 1990 Jul-Aug;3(4):247-51. doi: 10.1016/0920-9964(90)90005-r. PMID 2278986
- [Background] Sarróa S, Dueñasa R, Galvea L, Mediavillac R, Mensad I, Soléa J, et al. Validación de la escala de Calgary en pacientes con esquizofrenia crónica. Informaciones Psiquiátricas. 2005; 182: 203-214.
- [Background] Alonso J, Prieto L, Anto JM. [The Spanish version of the SF-36 Health Survey (the SF-36 health questionnaire): an instrument for measuring clinical results]. Med Clin (Barc). 1995 May 27;104(20):771-6. Spanish. PMID 7783470
- [Background] Dois A, Contreras A, Arechabala M, Urrutia S. Validación de una escala de calidad de vida en un grupo de personas con esquizofrenia en la Región Metropolitana- Chile. Cienc. enferm. 2007, 13(1): 35-44.
- [Background] Mattick RP, Clarke JC. Development and validation of measures of social phobia scrutiny fear and social interaction anxiety. Behav Res Ther. 1998 Apr;36(4):455-70. doi: 10.1016/s0005-7967(97)10031-6. PMID 9670605
- [Background] De la Rubia J, García C, Antona C. Validación de la escala de ansiedad en la interacción social en estudiantes universitarios mexicanos. Pensam. psicol. 2013. 11 (1): 27-42.
- [Background] Kennedy RS, Lane NE, Berbaum KS, Lilienthal MG. Simulator sickness questionnaire: an enhanced method for quantifying simulator sickness. Int. J. Aviat. Psychol. 1993; 3(3): 203-220.
- [Background] Bedregal P, Margozzini P, González C. Informe final estudio de carga de enfermedad y carga atribuible. Santiago de Chile: Ministerio de Salud, Gobierno de Chile; 2008.